CLINICAL TRIAL: NCT01972607
Title: The Effect of Aerobic Exercise Training for Migraine Prevention.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Collaborators: Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Responsible Party: Principal Investigator, Arão Belitardo de Oliveira, Prof. BS. Arão Belitardo de Oliveira, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 081511
Record Dates: First submitted 2013-10-21; First posted 2013-10-30 (Estimated); Last update posted 2020-12-29 (Actual); Status verified 2020-12

CONDITIONS: Headache Disorders, Primary
Keywords: Migraine, aerobic exercise, prevention
MeSH Terms: conditions — Headache Disorders, Primary; Migraine Disorders | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- CONTROL (No Intervention): This group will receive the same treatment of the experimental group after the test-retest measurements.
- EXERCISE (Experimental): This group will receive the treatment with aerobic exercise training
  Interventions: Other: Exercise Training

INTERVENTIONS:
Other: Exercise Training — 12 weeks of aerobic exercise training performed 3x/week at moderate intensity with sessions of 40 min.
  Arms: EXERCISE

SUMMARY:
This study has been designed in order to know the effect of 12 weeks of aerobic exercise training for migraine prevention. We hypothesized that the exercise training could reduce the number of days with migraine and the number of attacks per month in the treated group.

DETAILED DESCRIPTION:
The study will cover 20 weeks. The first 8 weeks has been designed as "baseline" period, to assess the migraine status and classification, colect blood exam, perform a cardiopulmonary exercise test to determine the maximal oxygen uptake, and fill psychometric questionnaires. The remaining 12 weeks will be the "intervention" period, where participants after randomization will be allocated to perform an aerobic exercise training (on treadmill) performed on a 3 times per week-based program of 40-min duration each session, or will wait for the equal period to repeat all the assessments, then begin the same exercise protocol.

ELIGIBILITY:
Inclusion Criteria:

* Sedentary (> 6 month) healthy subjects and sedentary (> 6 month)subjects with migraine without aura, migraine with aura and chronic migraine;

Exclusion Criteria:

* Physically active(> 1 day/week);
* Tobacco user;
* Alcohol or abuse drug user;
* Taking any prescribed medication or, in the case of medication for migraine prevention, if taking < 6 months.
* Having any cardiovascular, pulmonary, endocrine-metabolic, rheumatic or other neurologic disease or psychiatric disorder such as bipolar disorder and post-traumatic stress disorder.
* Undergoing surgical procedure less than 3 months before entering the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-03; Primary Completion 2015-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Frequency of Migraine/month | Migraine frequency measured between 4th and 8th weeks has been set as the "baseline" period, and will be compared to changes in frequency measured between weeks 12 to 16, which has been set as "post-intervention" period.
Plasma levels of anandamide, cytokines and aminopeptidases | Resting plasma levels measured between 4th and 8th weeks has been set as the "baseline" levels, and will be compared to changes in resting levels measured between weeks 12 to 16, set as the "post-intervention" levels.

SECONDARY OUTCOMES:
Days with Migraine | Days with migraine measured between 4th and 8th weeks has been set as the "baseline" period, and will be compared to changes in days with migraine measured between weeks 12 to 16, which has been set as "post-intervention" period

OTHER OUTCOMES:
Maximal Oxygen Uptake | Measurements of the maximal oxygen uptake has been performed at Week 1, which is set as "baseline" measurement, and at week 16, which is set as "post-intervention" measurement.

CONTACTS AND LOCATIONS:
Overall Officials: Mario FP Peres, MD, PhD, Study Chair — Federal University of São Paulo
Locations (1):
- Federal University of Sao Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Oliveira AB, Ribeiro RT, Mello MT, Tufik S, Peres MFP. Anandamide Is Related to Clinical and Cardiorespiratory Benefits of Aerobic Exercise Training in Migraine Patients: A Randomized Controlled Clinical Trial. Cannabis Cannabinoid Res. 2019 Dec 9;4(4):275-284. doi: 10.1089/can.2018.0057. eCollection 2019. PMID 31872062
- [Derived] Belitardo de Oliveira A, de Mello MT, Tufik S, Peres MFP. Weight loss and improved mood after aerobic exercise training are linked to lower plasma anandamide in healthy people. Physiol Behav. 2019 Mar 15;201:191-197. doi: 10.1016/j.physbeh.2018.12.018. Epub 2018 Dec 19. PMID 30578894